CLINICAL TRIAL: NCT00460525
Title: Randomized, Controlled Phase II Clinical Trial to Evaluate the Safety, Immunogenicity and Efficacy of the AMA-1 Malaria Vaccine FMP2.1/AS02A Versus Rabies Vaccine in 1-6 Year Old Children in Bandiagara, Mali
Brief Title: Phase II AMA-1 Malaria Vaccine FMP2.1/AS02A Trial in Mali
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); GlaxoSmithKline (Industry); University of Maryland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 07-0003; U01AI065683 (NIH); 2U01AI065683-06 (NIH); Malaria-056 (110060) (Other: GSK); HSRRB # A-14262 (Other: USAMRMC)
Record Dates: First submitted 2007-04-12; First posted 2007-04-16 (Estimated); Results first posted 2010-08-10 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Plasmodium Falciparum Malaria
Keywords: malaria, Mali, children, Plasmodium falciparum, vaccine
MeSH Terms: conditions — Malaria, Falciparum; Malaria | interventions — Rabies Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rabies Vaccine (Active Comparator): Rabies vaccine administered on Days 0, 30, and 60.
  Interventions: Biological: Rabies Vaccine
- FMP2.1/AS02A (Experimental): 50 mcg of FMP2.1 in 0.5 mL AS02A administered on Days 0, 30, and 60.
  Interventions: Biological: FMP2.1/AS02A

INTERVENTIONS:
Biological: FMP2.1/AS02A — 3 doses administered a month apart: 50 µg recombinant subunit protein FMP2.1 (Plasmodium falciparum Apical Membrane Antigen-1 from strain 3D7 expressed in and purified from Escherichia coli), adjuvanted with 0.5 mL of AS02A (proprietary oil-in-water emulsion and phosphate buffered saline with the immunostimulants monophosphoral lipid A and QS21).
  Arms: FMP2.1/AS02A
Biological: Rabies Vaccine — White, freeze-dried vaccine for reconstitution with the diluent prior to use; dosage 1.0 mL of rabies vaccine.
  Arms: Rabies Vaccine

SUMMARY:
Malaria is a disease that affects many people in Africa. Malaria is caused by germs spread by mosquito bites. The purpose of this study is to compare the number of children who get malaria after receiving an experimental malaria vaccine (FMP2.1/AS02A) to the number of children who get malaria after receiving a vaccine for rabies (an approved vaccine that does not prevent malaria). The children will be assigned to one of the vaccine groups by chance. Participants and doctors will not know which vaccine was given. Study participants will include 400 children, ages 1-6 years, living in Bandiagara, Mali. Children will receive 3 vaccine doses, by injection, to their upper arm. Study procedures will include physical exams and several blood samples. Participants will be involved in the study for 26 months.

DETAILED DESCRIPTION:
This is a randomized, controlled, phase II clinical trial to evaluate the efficacy, safety and immunogenicity of the apical membrane antigen-1 of Plasmodium (P.) falciparum (AMA-1) malaria vaccine FMP2.1/AS02A using rabies vaccine as a control in healthy children 1-6 years old in Bandiagara, Mali. This study is linked to DMID protocol 05-0146, which is a phase I dose escalation trial at the same site in the same population. In this study, 400 subjects will be randomized in a 1:1 ratio to receive either 50 micrograms of FMP2.1 in 0.5 mL AS02A or rabies vaccine. Immunizations will be given on days 0, 30 and 60. Solicited adverse events will be recorded on the days of immunization and at 1, 2, 3 and 7 days after each immunization. Unsolicited adverse events will be recorded for 30 days after each immunization. Passive case detection will be used to capture clinical malaria episodes and adverse events including serious adverse events, and will occur by continuous availability of clinical care in a population with high utilization of this care. Active surveillance will be used to capture malaria infections and adverse events including serious adverse events. For active case detection, following the third dose, participants will be followed monthly for 6 months and then at 12, 18 and 24 months after randomization, for clinical assessment, malaria smear and hemoglobin. Routine monthly malaria smears will not be read immediately unless symptoms are present. Children will be followed for 2 years after the first immunization. Sera will be collected for anti-FMP2.1 antibody titers on the days of immunization and 1, 3, 6, 8, 12, 18 and 24 months after the first immunization. Peripheral blood mononuclear cells (PBMCs) will be collected on the days of immunization, 30 days after the third immunization and 8, 12, 18 and 24 months after the first immunization. The study Final Report will be based on data collected up to 6 months after the assigned date of the third immunization. A supplemental report will include data from the entire 24-month observation period. Primary study objectives are to: determine the efficacy of FMP2.1/AS02A in children aged 1-6 years against first clinical malaria episodes (axillary temperature of greater than or equal to 37.5 degrees Celsius and parasitemia of greater than or equal to 2500/mm^3) occurring between randomization and 6 months after the assigned date of the third immunization; and assess the safety of the vaccine in children aged 1-6 years. Secondary study objectives are to: describe the dynamics of anti-AMA-1 antibody responses in recipients of the malaria vaccine compared to natural responses in the control group; determine whether serum anti-AMA-1 IgG titer by enzyme linked immunosorbent assay (ELISA) 1 month after the third immunization correlates with protection against clinical malaria episode; measure allele-specific efficacy against parasites with AMA-1 genotypes homologous to and heterologous to the 3D7 clone of P. falciparum; determine vaccine efficacy against clinical malaria episodes occurring between randomization and 6 months after the assigned date of the third immunization; and if efficacy is observed based on the primary endpoint, to determine vaccine efficacy against first clinical malaria episode and all clinical episodes (using increasing parasitemia thresholds) occurring during 2 years after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-6 years inclusive at the time of screening
* Residing in Bandiagara town
* Appear to be in generally good health based on clinical and laboratory investigation
* Separate written informed consent obtained from the parent/guardian before screening and study start, respectively
* Available to participate in follow-up for the duration of study (26 months)

Exclusion Criteria:

* Previous vaccination with an investigational vaccine or a rabies vaccine
* Use of an investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first study immunization, or planned use up to 30 days after the third immunization
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first immunization. This exclusion includes any dose level of oral steroids or inhaled steroids, but not topical steroids.
* Confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection
* Confirmed or suspected autoimmune disease
* History of allergic reactions or anaphylaxis to immunizations or to any vaccine component
* History of serious allergic reactions to any substance, requiring hospitalization or emergent medical care
* History of allergy to tetracycline, doxycycline, nickel, Imidazole, eggs, neomycin, chlortetracycline or amphotericin B
* History of splenectomy
* Laboratory evidence of liver disease (alanine aminotransferase [ALT] greater than the upper limit of normal of the testing laboratory = 49.6 U/L)
* Laboratory evidence of renal disease (serum or plasma creatinine greater than 62 micro mol/L), or more than trace protein or blood on urine dipstick testing)
* Laboratory evidence of hematologic disease (absolute leukocyte count <5,300/mm^3 or >15,300/mm^3, absolute lymphocyte count <2,300 mm^3, platelet count <133,000/mm^3, or hemoglobin <9.0 g/dL)
* Hepatitis B surface antigen positive
* Chronic skin condition that could interfere with vaccine site reactogenicity assessment
* Administration of immunoglobulins and/or any blood products within the three months preceding the first study immunization or planned administration during the study period
* Simultaneous participation in any other interventional clinical trial
* Acute or chronic pulmonary, cardiovascular, hepatic (including hepatomegaly), renal or neurological condition, severe malnutrition, or any other clinical findings that in the opinion of the PI may increase the risk of participating in the study
* Other condition that in the opinion of the Principal Investigator (PI) would jeopardize the safety or rights of a participant in the trial or would render the participant unable to comply with the protocol

Ages: 1 Year to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 400 (Actual)
Dates: Start 2007-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mahamadou A Thera, MD, MPH, Principal Investigator — University of Bamako
Locations (1):
- University of Bamako, Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Result] Dutta S, Lalitha PV, Ware LA, Barbosa A, Moch JK, Vassell MA, Fileta BB, Kitov S, Kolodny N, Heppner DG, Haynes JD, Lanar DE. Purification, characterization, and immunogenicity of the refolded ectodomain of the Plasmodium falciparum apical membrane antigen 1 expressed in Escherichia coli. Infect Immun. 2002 Jun;70(6):3101-10. doi: 10.1128/IAI.70.6.3101-3110.2002. PMID 12011004
- [Result] Polhemus ME, Magill AJ, Cummings JF, Kester KE, Ockenhouse CF, Lanar DE, Dutta S, Barbosa A, Soisson L, Diggs CL, Robinson SA, Haynes JD, Stewart VA, Ware LA, Brando C, Krzych U, Bowden RA, Cohen JD, Dubois MC, Ofori-Anyinam O, De-Kock E, Ballou WR, Heppner DG Jr. Phase I dose escalation safety and immunogenicity trial of Plasmodium falciparum apical membrane protein (AMA-1) FMP2.1, adjuvanted with AS02A, in malaria-naive adults at the Walter Reed Army Institute of Research. Vaccine. 2007 May 22;25(21):4203-12. doi: 10.1016/j.vaccine.2007.03.012. Epub 2007 Mar 26. PMID 17442466
- [Derived] Laurens MB, Kouriba B, Bergmann-Leitner E, Angov E, Coulibaly D, Diarra I, Daou M, Niangaly A, Blackwelder WC, Wu Y, Cohen J, Ballou WR, Vekemans J, Lanar DE, Dutta S, Diggs C, Soisson L, Heppner DG, Doumbo OK, Plowe CV, Thera MA. Strain-specific Plasmodium falciparum growth inhibition among Malian children immunized with a blood-stage malaria vaccine. PLoS One. 2017 Mar 10;12(3):e0173294. doi: 10.1371/journal.pone.0173294. eCollection 2017. PMID 28282396
- [Derived] Graves SF, Kouriba B, Diarra I, Daou M, Niangaly A, Coulibaly D, Keita Y, Laurens MB, Berry AA, Vekemans J, Ripley Ballou W, Lanar DE, Dutta S, Gray Heppner D, Soisson L, Diggs CL, Thera MA, Doumbo OK, Plowe CV, Sztein MB, Lyke KE. Strain-specific Plasmodium falciparum multifunctional CD4(+) T cell cytokine expression in Malian children immunized with the FMP2.1/AS02A vaccine candidate. Vaccine. 2016 May 17;34(23):2546-55. doi: 10.1016/j.vaccine.2016.04.019. Epub 2016 Apr 15. PMID 27087149
- [Derived] Laurens MB, Thera MA, Coulibaly D, Ouattara A, Kone AK, Guindo AB, Traore K, Traore I, Kouriba B, Diallo DA, Diarra I, Daou M, Dolo A, Tolo Y, Sissoko MS, Niangaly A, Sissoko M, Takala-Harrison S, Lyke KE, Wu Y, Blackwelder WC, Godeaux O, Vekemans J, Dubois MC, Ballou WR, Cohen J, Dube T, Soisson L, Diggs CL, House B, Bennett JW, Lanar DE, Dutta S, Heppner DG, Plowe CV, Doumbo OK. Extended safety, immunogenicity and efficacy of a blood-stage malaria vaccine in malian children: 24-month follow-up of a randomized, double-blinded phase 2 trial. PLoS One. 2013 Nov 18;8(11):e79323. doi: 10.1371/journal.pone.0079323. eCollection 2013. PMID 24260195
- [Derived] Thera MA, Doumbo OK, Coulibaly D, Laurens MB, Ouattara A, Kone AK, Guindo AB, Traore K, Traore I, Kouriba B, Diallo DA, Diarra I, Daou M, Dolo A, Tolo Y, Sissoko MS, Niangaly A, Sissoko M, Takala-Harrison S, Lyke KE, Wu Y, Blackwelder WC, Godeaux O, Vekemans J, Dubois MC, Ballou WR, Cohen J, Thompson D, Dube T, Soisson L, Diggs CL, House B, Lanar DE, Dutta S, Heppner DG Jr, Plowe CV. A field trial to assess a blood-stage malaria vaccine. N Engl J Med. 2011 Sep 15;365(11):1004-13. doi: 10.1056/NEJMoa1008115. PMID 21916638

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the population of healthy children aged 1-6 years residing in the town of Bandiagara.
Period: Overall Study
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Started | 201 | 199
Completed | 190 | 194
Not Completed | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabies Vaccine | FMP2.1/AS02A | Total
Number analyzed (Participants) | 201 | 199 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 201 | 199 | 400
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.4 (1.5) | 3.4 (1.6) | 3.4 (1.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 103 | 215
  Male | 89 | 96 | 185
Region of Enrollment [Number; unit: participants]
  Mali | 201 | 199 | 400

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events During the 7-day Surveillance Period After the First Vaccination
Description: Solicited symptoms were recorded by study staff at clinic visits on Days 0, 1, 2 and 7 after each vaccination. "Reported Limitation of Arm Motion" refers to the parents' report of the symptom while "Limitation of Arm Motion" refers to the clinicians' assessment of the symptom, collected separately.
Time Frame: 0-7 days after first vaccination
Population: All subjects receiving the vaccination are included.
Measure: Number; unit: Participants
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 201 | 199
Participants
  Drowsiness | 0 | 5
  Irritability/Fussiness | 0 | 12
  Loss of Appetite | 3 | 25
  Vomiting | 1 | 4
  Fever | 30 | 61
  Site Pain | 55 | 157
  Swelling | 34 | 153
  Erythema | 0 | 12
  Reported Limitation of Arm Motion | 4 | 55
  Limitation of Arm Motion | 2 | 54

2. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events During the 7-day Surveillance Period After the Second Vaccination.
Description: Solicited symptoms were recorded by study staff at clinic visits on Days 0, 1, 2 and 7 after vaccination. "Reported Limitation of Arm Motion" refers to the parents' report of the symptom while "Limitation of Arm Motion" refers to the clinicians' assessment of the symptom, collected separately.
Time Frame: 0-7 days after the second vaccination
Population: All subjects receiving the vaccination are included.
Measure: Number; unit: Participants
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 193 | 193
Participants
  Drowsiness | 0 | 0
  Irritability/Fussiness | 1 | 5
  Loss of Appetite | 1 | 10
  Vomiting | 3 | 3
  Fever | 13 | 64
  Site Pain | 57 | 132
  Swelling | 69 | 151
  Erythema | 0 | 1
  Reported Limitation of Arm Motion | 0 | 31
  Limitation of Arm Motion | 2 | 37

3. Primary Outcome: Number of Subjects Reporting Solicited Adverse Events During the 7-day Surveillance Period After the Third Vaccination.
Description: as for outcome 2
Time Frame: 0-7 days after the third vaccination
Population: All subjects receiving the vaccination are included.
Measure: Number; unit: Participants
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 187 | 184
Participants
  Drowsiness | 1 | 0
  Irritability/Fussiness | 2 | 6
  Loss of Appetite Post | 0 | 3
  Vomiting | 2 | 2
  Fever | 18 | 64
  Site Pain | 48 | 134
  Swelling | 90 | 159
  Erythema | 0 | 3
  Reported Limitation of Arm Motion | 4 | 26
  Limitation of Arm Motion | 2 | 28

4. Primary Outcome: Number of Unsolicited Non-serious Adverse Events Reported During the 30-day Surveillance Period After the First Vaccination
Description: Unsolicited non-serious adverse events reported are those occurring within 30 days after vaccination. The categories are the MedDRA System Organ Classes for which at least one adverse event was reported. All non-serious adverse events are included, regardless of severity or relationship to vaccination.
Time Frame: Day 0-29 after first vaccination
Population: All subjects receiving the vaccination are included.
Measure: Number; unit: Adverse Events
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 201 | 199
Adverse Events
  Blood and lymphatic system disorders | 7 | 4
  Ear and labyrinth disorders | 0 | 0
  Eye disorders | 5 | 5
  Gastrointestinal disorders | 17 | 11
  General disorders, administrative site conditions | 16 | 44
  Hepatobiliary disorders | 2 | 0
  Infections and infestations | 56 | 53
  Injury, poisoning, and procedural complications | 5 | 4
  Investigations | 45 | 42
  Metabolism and nutrition disorders | 0 | 0
  Musculoskeletal and connective tissue disorders | 0 | 0
  Nervous system disorders | 3 | 2
  Psychiatric disorders | 0 | 4
  Renal and urinary disorders | 1 | 1
  Reproductive system and breast disorders | 1 | 2
  Respiratory, thoracic and mediastinal disorders | 23 | 28
  Skin and subcutaneous tissue disorders | 5 | 6
  Vascular disorders | 0 | 0

5. Primary Outcome: Number of Unsolicited Non-serious Adverse Events Reported During the 30-day Surveillance Period After the Second Vaccination
Description: as for outcome 4
Time Frame: Day 0-29 after second vaccination
Population: All subjects receiving the vaccination are included.
Measure: Number; unit: Adverse Events
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 193 | 193
Adverse Events
  Blood and lymphatic system disorders | 1 | 2
  Ear and labyrinth disorders | 0 | 1
  Eye disorders | 1 | 1
  Gastrointestinal disorders | 19 | 11
  General disorders, administrative site conditions | 9 | 26
  Hepatobiliary disorders | 0 | 0
  Infections and infestations | 67 | 68
  Injury, poisoning, and procedural complications | 6 | 3
  Investigations | 71 | 74
  Metabolism and nutrition disorders | 0 | 1
  Musculoskeletal and connective tissue disorders | 0 | 1
  Nervous system disorders | 0 | 1
  Psychiatric disorders | 1 | 1
  Renal and urinary disorders | 0 | 1
  Reproductive system and breast disorders | 0 | 1
  Respiratory, thoracic and mediastinal disorders | 17 | 16
  Skin and subcutaneous tissue disorders | 4 | 5
  Vascular disorders | 0 | 0

6. Primary Outcome: Number of Unsolicited Non-serious Adverse Events Reported During the 30-day Surveillance Period After the Third Vaccination
Description: as for outcome 4
Time Frame: Day 0-29 after third vaccination
Population: All subjects receiving the vaccination are included.
Measure: Number; unit: Adverse Events
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 187 | 184
Adverse Events
  Blood and lymphatic system disorders | 7 | 1
  Ear and labyrinth disorders | 0 | 0
  Eye disorders | 8 | 7
  Gastrointestinal disorders | 13 | 16
  General disorders, administrative site conditions | 14 | 29
  Hepatobiliary disorders | 0 | 0
  Infections and infestations | 84 | 73
  Injury, poisoning, and procedural complications | 6 | 5
  Investigations | 110 | 109
  Metabolism and nutrition disorders | 2 | 0
  Musculoskeletal and connective tissue disorders | 0 | 0
  Nervous system disorders | 5 | 1
  Psychiatric disorders | 1 | 1
  Renal and urinary disorders | 0 | 0
  Reproductive system and breast disorders | 0 | 0
  Respiratory, thoracic and mediastinal disorders | 32 | 36
  Skin and subcutaneous tissue disorders | 7 | 9
  Vascular disorders | 0 | 1

7. Primary Outcome: Time to First Clinical Malaria Episode With Significant Parasitemia (2500/mm^3) and Temperature of Greater Than or Equal to 37.5 Degrees C.
Description: Time to first clinical malaria episode is displayed in a life table format to display the number of subjects at risk, the number with first clinical episode and the number censored at each time point.
Time Frame: Occurring between randomization and 6 months after the assigned date of the 3rd immunization.
Measure: Number; unit: Participants
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 201 | 199
Participants
  Days 0 - 30, Number at Risk | 201 | 199
  Days 0 - 30, Number with First Episode | 1 | 0
  Days 0 -30, Number Censored | 4 | 1
  Days 31 - 60, Number at Risk | 196 | 198
  Days 31 - 60, Number with First Episode | 9 | 10
  Days 31 - 60, Number Censored | 1 | 0
  Days 61 - 90 Number at Risk | 186 | 188
  Days 61 - 90, Number with First Episode | 40 | 25
  Days 61 - 90, Number Censored | 0 | 1
  Days 91 - 120, Number at Risk | 146 | 162
  Days 91 - 120, Number with First Episode | 28 | 33
  Days 91 - 120, Number Censored | 0 | 0
  Days 121 - 150, Number at Risk | 118 | 129
  Days 121 - 150, Number with First Episode | 16 | 10
  Days 121 - 150, Number Censored | 1 | 1
  Days 151 - 180, Number at Risk | 101 | 118
  Days 151 - 180, Number with First Episode | 5 | 9
  Days 151 - 180, Number Censored | 2 | 1
  Days 181 - 210, Number at Risk | 94 | 108
  Days 181 - 210, Number with First Episode | 5 | 5
  Days 181 - 210, Number Censored | 0 | 0
  Days 211 - 240, Number at Risk | 89 | 103
  Days 211 - 240, Number with First Episode | 2 | 3
  Days 211 - 240, Number Censored | 87 | 100
Statistical Analysis 1: Comparison: Rabies Vaccine vs FMP2.1/AS02A; Time to first clinical malaria episode with significant parasitemia (2500/mm^3) and temperature of greater than or equal to 37.5 degrees C was analyzed by fitting a Cox Proportional Hazards model. The null hypothesis of no vaccine efficacy was tested by the stratified log-rank test (score test). The point and interval estimates for vaccine efficacy were obtained by transforming those for treatment effect in the model; Test type: Superiority or Other; p = 0.175, Regression, Cox — The a priori threshold for statistical significance was set at 0.05; No adjustments were made; Vaccine Efficacy, VE=1-RR=1-exp(ß) = 0.17, 95% CI [-0.09 to 0.37] — Vaccine efficacy (VE) was defined as one minus the relative risk (RR), which was estimated by exponentiating the treatment parameter (ß) from the Cox model fit

8. Primary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: A serious adverse event was defined as any untoward medical occurrence that results in death, is life threatening, results in persistent or significant disability/incapacity, requires in-patient hospitalization or prolongation of existing hospitalization or is a congenital anomaly/birth defect in the offspring of a study subject. In addition, important medical events that may jeopardize the participant or may require intervention to prevent one of the other outcomes listed above was considered serious.
Time Frame: 24 months after initial vaccination
Measure: Number; unit: Participants
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 201 | 199
Participants | 2 | 8

9. Secondary Outcome: Incidence Density of Clinical Malaria Episode
Description: Clinical malaria episode was defined by significant parasitemia (2500/mm^3) and temperature of greater than or equal to 37.5 degrees C. Event rate was determined by dividing the number of episodes (150 for the Rabies group and 121 for the FMP2.1/ASO2A group) by the number of Person Years at Risk (PYAR) (126.341 for Rabies group and 127.411 for the FMP2.1/ASO2A group).
Time Frame: Between randomization and 6 months after 3rd immunization.
Population: Analyses are ITT.
Measure: Number; unit: Events Per PYAR
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 201 | 199
Events Per PYAR | 1.187263 | 0.949683
Statistical Analysis 1: Comparison: Rabies Vaccine vs FMP2.1/AS02A; Incidence density, defined as number of clinical malaria episodes per PYAR, was compared using Poisson regression. The null hypothesis of no vaccine efficacy was tested. The point and interval estimates for vaccine efficacy were obtained by transforming those for treatment effect in the model; Test type: Superiority or Other; p = 0.068, Poisson regression — The a priori threshold for statistical significance was set at 0.05; No adjustments; Vaccine Efficacy, VE=1-RR=1-exp(ß) = 0.20, 95% CI [-0.02 to 0.37] — Vaccine efficacy (VE) was defined as one minus the relative risk (RR), which was estimated by exponentiating the treatment parameter (ß) from the Poisson model fit

10. Secondary Outcome: Geometric Mean Titers of Anti-FMP2.1 Antibody Measured by Enzyme Linked ImmunoSorbent Assay (ELISA) at Day 0
Description: Titers of Anti-FMP2.1 antibody were determined by ELISA from sera collected at Day 0 prior to the first vaccination.
Time Frame: Day 0
Population: Analyses are ITT. No imputation techniques were used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 201 | 199
Titer | 430.4 [298.0 to 621.4] | 393.1 [273.2 to 565.5]

11. Secondary Outcome: Geometric Mean Titers of Anti-FMP2.1 Antibody Measured by ELISA at Day 30.
Description: Titers of Anti-FMP2.1 antibody were determined by ELISA from sera collected at Day 30, prior to the second vaccination.
Time Frame: Day 30 after initial vaccination
Population: Analyses are ITT. No imputation techniques were used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 195 | 194
Titer | 403.7 [275.8 to 591.0] | 21248.7 [17616.8 to 25629.5]

12. Secondary Outcome: Geometric Mean Titers of Anti-FMP2.1 Antibody Measured by ELISA at Day 60.
Description: Titers of Anti-FMP2.1 antibody were determined by ELISA from sera collected at Day 60, prior to the third vaccination.
Time Frame: Day 60 after initial vaccination
Population: Analyses are ITT. No imputation techniques were used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 194 | 195
Titer | 512.2 [350.1 to 749.3] | 98199.0 [86574.6 to 111384.1]

13. Secondary Outcome: Geometric Mean Titers of Anti-FMP2.1 Antibody Measured by ELISA at Day 90.
Description: Titers of Anti-FMP2.1 antibody were determined by ELISA from sera collected at Day 90.
Time Frame: Day 90 after initial vaccination
Population: Analyses are ITT. No imputation techniques were used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 191 | 194
Titer | 781.8 [524.8 to 1164.5] | 188449.1 [165625.5 to 214417.8]

14. Secondary Outcome: Geometric Mean Titers of Anti-FMP2.1 Antibody Measured by ELISA at Day 150.
Description: Titers of Anti-FMP2.1 antibody were determined by ELISA from sera collected at Day 150.
Time Frame: Day 150 after initial vaccination
Population: Analyses are ITT. No imputation techniques were used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 188 | 194
Titer | 1202.9 [813.3 to 1779.0] | 100746.5 [85163.0 to 119181.5]

15. Secondary Outcome: Geometric Mean Titers of Anti-FMP2.1 Antibody Measured by ELISA at Day 240.
Description: Titers of Anti-FMP2.1 antibody were determined by ELISA from sera collected at Day 240.
Time Frame: Day 240 after initial vaccination
Population: Analyses are ITT. No imputation techniques were used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 189 | 193
Titer | 774.6 [525.5 to 1141.8] | 65031.7 [54999.2 to 76894.4]

16. Secondary Outcome: Geometric Mean Titers of Anti-FMP2.1 Antibody Measured by ELISA at Day 364
Description: Titers of Anti-FMP2.1 antibody were determined by ELISA from sera collected at Day 364.
Time Frame: Day 364 after initial vaccination
Population: Analyses are ITT. No imputation techniques were used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 185 | 192
Titer | 505.0 [353.9 to 720.5] | 42596.8 [36549.9 to 49644.1]

17. Secondary Outcome: Geometric Mean Titers of Anti-FMP2.1 Antibody Measured by ELISA at Day 547
Description: Titers of Anti-FMP2.1 antibody were determined by ELISA from sera collected at Day 547.
Time Frame: Day 547 after initial vaccination
Population: Analyses are ITT. No imputation techniques were used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 183 | 183
Titer | 1589.3 [1075.0 to 2349.7] | 81205.1 [66166.2 to 99662.1]

18. Secondary Outcome: Geometric Mean Titers of Anti-FMP2.1 Antibody Measured by ELISA at Day 730
Description: Titers of Anti-FMP2.1 antibody were determined by ELISA from sera collected at Day 730.
Time Frame: Day 730 after initial vaccination
Population: Analyses are ITT. No imputation techniques were used.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Number analyzed (Participants) | 168 | 179
Titer | 636.5 [431.4 to 939.0] | 40605.3 [33946.8 to 48569.8]

ADVERSE EVENTS:
Time Frame: Solicited adverse events were collected for 7 days after each immunization. Serious adverse events and unsolicited non-serious adverse events were collected for 24 months after initial vaccination.
Arm/Group | Rabies Vaccine | FMP2.1/AS02A
Serious Adverse Events (participants affected / at risk) | 2/201 | 8/199
Other Adverse Events (participants affected / at risk) | 198/201 | 199/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rabies Vaccine (N=201) | FMP2.1/AS02A (N=199)
Malaria (Infections and infestations) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Febrile Convulsion (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral malaria (Infections and infestations) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rabies Vaccine (N=201) | FMP2.1/AS02A (N=199)
Conjunctivitis (Eye disorders) | 55 (71) | 49 (61)
Abdominal Pain (Gastrointestinal disorders) | 39 (57) | 45 (74)
Diarrhoea (Gastrointestinal disorders) | 64 (96) | 48 (81)
Vomiting (Gastrointestinal disorders) | 17 (20) | 24 (30)
Pyrexia (General disorders) | 50 (65) | 89 (120)
Bronchitis (Infections and infestations) | 126 (273) | 121 (259)
Ear infection (Infections and infestations) | 47 (65) | 46 (55)
Fungal skin infection (Infections and infestations) | 27 (31) | 24 (27)
Furuncle (Infections and infestations) | 18 (18) | 17 (20)
Mumps (Infections and infestations) | 19 (19) | 12 (12)
Nasopharyngitis (Infections and infestations) | 43 (59) | 41 (54)
Pharyngitis (Infections and infestations) | 31 (32) | 33 (40)
Pneumonia (Infections and infestations) | 31 (37) | 33 (42)
Pyoderma (Infections and infestations) | 54 (71) | 60 (89)
Rhinitis (Infections and infestations) | 127 (244) | 123 (251)
Salmonellosis (Infections and infestations) | 11 (13) | 5 (5)
Staphylococcal infection (Infections and infestations) | 12 (12) | 11 (11)
Tinea capitis (Infections and infestations) | 30 (36) | 26 (27)
Tonsillitis (Infections and infestations) | 19 (22) | 18 (22)
Trichomoniasis intestinal (Infections and infestations) | 12 (13) | 19 (21)
Varicella (Infections and infestations) | 57 (57) | 49 (50)
Wound (Injury, poisoning and procedural complications) | 39 (51) | 41 (49)
Alanine aminotransferase increased (Investigations) | 12 (13) | 10 (11)
Granulocyte count increased (Investigations) | 36 (37) | 24 (24)
Haemoglobin increased (Investigations) | 94 (145) | 92 (143)
Lymphocyte count decreased (Investigations) | 12 (12) | 13 (14)
Lymphocyte count increased (Investigations) | 10 (12) | 16 (16)
Platelet count increased (Investigations) | 47 (60) | 59 (80)
Red blood cell count increased (Investigations) | 15 (16) | 4 (5)
White blood cell count decreased (Investigations) | 18 (21) | 17 (19)
White blood cell count increased (Investigations) | 17 (19) | 18 (19)
Anorexia (Metabolism and nutrition disorders) | 11 (11) | 4 (4)
Headache (Nervous system disorders) | 25 (34) | 30 (36)
Cough (Respiratory, thoracic and mediastinal disorders) | 109 (166) | 104 (190)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 39 (46) | 28 (30)
Rash papular (Skin and subcutaneous tissue disorders) | 7 (8) | 11 (13)
Skin lesion (Skin and subcutaneous tissue disorders) | 6 (8) | 11 (11)
Injection site erythema (General disorders) | 0 (0) | 13 (13)
Injection site pain (General disorders) | 92 (114) | 180 (324)
Injection site swelling (General disorders) | 129 (167) | 192 (438)
Irritability (General disorders) | 1 (1) | 17 (19)
Pyrexia (General disorders) | 46 (52) | 104 (133)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 32 (35)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less